CLINICAL TRIAL: NCT02803593
Title: To Enhance Breast Cancer Survivorship of Asian Americans
Acronym: TICAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eun-Ok Im, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00117270; R01CA203719-01 (NIH)
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: technology-based intervention; Asian American; survivorship
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Asian American breast cancer survivors who do not use the TICAA, but use the information on breast cancer by the American Cancer Society (ACS). Participants are asked to use the online ACS resources for 3 months.
  Interventions: Behavioral: American Cancer Society information on breast cancer
- TICAA Intervention (Experimental): Asian American breast cancer survivors who use the TICAA intervention and the information by the ACS. The intervention is a technology-based information and coaching/support program to enhance survivorship experience of Asian American breast cancer survivors. Participants are asked to use the TICAA program for 3 months.
  Interventions: Behavioral: Technology-based information and coaching/support program; Behavioral: American Cancer Society information on breast cancer

INTERVENTIONS:
Behavioral: Technology-based information and coaching/support program — The TICAA has three components in four languages (English, Mandarin Chinese, Korean, and Japanese): (a) social media sites; (b) interactive online educational sessions; and (c) online resources. The social media sites provide a mechanism by which participants can receive coaching/support from culturally matched peers and health care providers. The educational sessions provide information about general and sub-ethnic- specific topics related to breast cancer survivorship. The online resources include 35 Web links to resources related to breast cancer survivorship from scientific authorities and from general and sub-ethnic-specific health organizations/institutes.
  Other Names: TICAA
  Arms: TICAA Intervention
Behavioral: American Cancer Society information on breast cancer — The American Cancer Society (ACS) webpage has a wide range of information on breast cancer including prevention, treatment, and ways to connect with breast cancer survivors.

SUMMARY:
The purpose of this randomized intervention study is to test the efficacy of the technology-based information and coaching/support program for Asian American breast cancer survivors (TICAA) in enhancing the women's breast cancer survivorship experience.

DETAILED DESCRIPTION:
Despite few studies on Asian American breast cancer survivors, it is well known that these women shoulder unnecessary burden of breast cancer because they rarely complain about symptoms or pain, delay seeking help, and rarely ask or get support due to their cultural values and beliefs and language barriers. This demonstrates a definite need for support in this specific population. However, survivorship programs that are increasingly instituted at cancer centers have serious impediments to providing information and coaching/support because of the lack of staff time and insurance reimbursement. Furthermore, the pressure of fast-paced clinical patient-provider interactions leaves little time for health care providers to provide up-to-date information and coaching or support for these women based on their cultural attitudes. All these circumstances necessitate an innovative and creative delivery method of information and coaching/support. A technology-based approach using computers and mobile devices (smart phones and tablets) promises to meet this necessity with high flexibility and accessibility, and minimizes the cost of the intervention in busy and costly health care settings. Also, a technology-based intervention that does not involve face-to-face interactions could work better for many women from cultures where breast cancer is still a stigmatizing experience. Therefore, based on preliminary studies, the research team has developed and pilot-tested a theory-driven technology-based information and coaching/support program that is culturally tailored to Asian American breast cancer survivors using multiple features. The purpose of the proposed randomized intervention study is to test the efficacy of the technology-based information and coaching/support program for Asian American breast cancer survivors (TICAA) in enhancing the women's breast cancer survivorship experience. The specific aims are to: a) determine whether the intervention group will show significantly greater improvements than the control group in primary outcomes (needs for help, physical and psychological symptoms, and quality of life) from baseline (pre-test) to Time Points 1 (post 1-month) and 2 (post 3-months); b) identify theory-based variables (attitudes, self-efficacy, perceived barriers, and social influences related to breast cancer survivorship) that mediate the intervention effects of the TICAA on the primary outcomes at the three time points (pre-test, post 1-month and post 3-months); and c) determine whether the effects of the TICAA on the primary outcomes are moderated by background characteristics and disease factors. The proposed study will be guided by the Bandura's Theory of Behavioral Change. This study adopts a randomized repeated measures pretest/posttest control group design in 330 Asian American breast cancer survivors. The long-term goals are to: (a) implement the program into various health care settings; (b) determine if the TICAA will lead to long-term improved health outcomes; and (c) fundamentally enhance the methodology/paradigm of culturally tailored technology-based interventions for ethnic minority groups of breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Asian American women aged 21 years and older who identify their sub-ethnicity as Chinese, Korean, or Japanese
* Have had a breast cancer diagnosis
* Can read and write English, Mandarin Chinese, Korean or Japanese
* Have access to the Internet through computers or mobile devices (smart phones and tablets)

Exclusion Criteria:

* Those under 21 years old are excluded because their cancer experience would be different from adults

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Ok Im, PhD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Duke University, School of Nursing, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Im EO, Chee W, Paul S, Kim SY, Choi MY, Mao JJ, Nguyen GT, Schapira MM, Ulrich CM, Yeo S, Deatrick JA, Inouye J, Ma G, Meghani S, Shin D, Bao T. Multiple dimensions of the quality of life among Asian American breast cancer survivors: The impact of a technology-based program. Breast. 2025 Aug;82:104490. doi: 10.1016/j.breast.2025.104490. Epub 2025 May 8. PMID 40359896
- [Derived] Im EO, Chee W, Paul S, Choi MY, Kim SY, Deatrick JA, Inouye J, Ma G, Meghani S, Nguyen GT, Schapira MM, Ulrich CM, Yeo S, Bao T, Shin D, Mao JJ. A randomized controlled trial testing a virtual program for Asian American women breast cancer survivors. Nat Commun. 2023 Oct 14;14(1):6475. doi: 10.1038/s41467-023-42132-6. PMID 37838727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Duke University in Durham, North Carolina, USA, and Emory University in Atlanta, Georgia, USA. Participant enrollment began in June 2016 and all follow up was complete by June 9, 2021.
Groups:
- Control: Asian American breast cancer survivors randomized to use the information on breast cancer by the American Cancer Society (ACS). Participants were asked to use the online ACS resources for 3 months.
- TICAA: Asian American breast cancer survivors randomized to use the TICAA intervention and the information by the ACS. The intervention is a technology-based information and coaching/support program to enhance survivorship experience of Asian American breast cancer survivors. Participants were asked to use the TICAA program for 3 months.
Period: Overall Study
Arm/Group | Control | TICAA
Started | 95 | 104
Completed Month 1 Assessment | 83 | 76
Completed (Completed the Month 3 assessment) | 78 | 69
Not Completed | 17 | 35
Not completed — Lost to Follow-up | 17 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | TICAA | Total
Number analyzed (Participants) | 95 | 104 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Some participants did not provide their age.
  years
    number analyzed (Participants) | 93 | 98 | 191
    (all) | 53.14 (13.62) | 51.60 (11.38) | 52.35 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 104 | 199
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 95 | 104 | 199
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 95 | 104 | 199
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self-identified ethnicity: Chinese | 52 | 36 | 88
  Self-identified ethnicity: Korean | 12 | 26 | 38
  Self-identified ethnicity: Japanese | 29 | 40 | 69
  Self-identified ethnicity: Not reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 95 | 104 | 199
Education [Count of Participants; unit: Participants]
  High school graduation or less | 33 | 21 | 54
  Completed undergraduate degree | 47 | 62 | 109
  Completed graduate degree | 15 | 21 | 36
Religion [Count of Participants; unit: Participants]
  No religion | 42 | 47 | 89
  Christian | 36 | 44 | 80
  Other | 16 | 13 | 29
  Not reported | 1 | 0 | 1
Marital status [Count of Participants; unit: Participants]
  Married, partnered, or in a permanent relationship | 70 | 73 | 143
  Single, divorced, or widowed | 25 | 30 | 55
  Not reported | 0 | 1 | 1
Employment status [Count of Participants; unit: Participants]
  Not employed | 52 | 55 | 107
  Employed | 34 | 38 | 72
  Not reported | 9 | 11 | 20
Birthplace [Count of Participants; unit: Participants]
  United States | 14 | 10 | 24
  Other than United States | 79 | 94 | 173
  Not reported | 2 | 0 | 2
Mean years living in United States [Mean (Standard Deviation); unit: years] — Population: Years living in the United States was determined for participants who were born outside of the United States.
  years
    number analyzed (Participants) | 79 | 94 | 173
    (all) | 18.73 (12.61) | 19.01 (11.42) | 18.88 (11.95)
Age at immigration [Mean (Standard Deviation); unit: years] — Population: Age at immigration was determined for participants who were born outside of the United States.
  years
    number analyzed (Participants) | 79 | 94 | 173
    (all) | 36.92 (12.32) | 32.33 (12.53) | 34.46 (12.60)
Acculturation score [Mean (Standard Deviation); unit: score on a scale] — The Suinn-Lew Asian Self Identity Acculturation Scale was administered to participants who were not born in the United States. This instrument assesses degree of acculturation with 21 items which are responded to on a 5-point scale. The final score is the average of responses to all items and ranges from 1 to 5 where 1 = low acculturation and 5 = high acculturation. Population: This assessment was administered to participants who were born outside of the United States.
  score on a scale
    number analyzed (Participants) | 79 | 94 | 173
    (all) | 3.55 (0.87) | 3.50 (0.74) | 3.52 (0.80)
Years since diagnosis [Mean (Standard Deviation); unit: years] | 3.73 (4.05) | 3.58 (3.74) | 3.65 (3.88)
Breast cancer type [Count of Participants; unit: Participants]
  Invasive | 56 | 71 | 127
  Non-invasive | 28 | 27 | 55
  Not reported | 11 | 6 | 17
Breast cancer stage [Count of Participants; unit: Participants] — Breast cancer staging describes how much cancer is present in the body, with higher stages indicating larger tumors and/or greater spread of cancer. Stage I describes a small, invasive tumor that has not spread to lymph nodes. Stages II and III describe tumors of increasing size with possible spread to axillary or mammary lymph nodes. Stage IV describes metastatic cancer that has spread to other organs, regardless of tumor size.
  Participants
    Stage I | 41 | 42 | 83
    Stage II/III | 40 | 51 | 91
    Stage IV | 4 | 4 | 8
    Unknown | 6 | 5 | 11
    Not reported | 4 | 2 | 6
Medical treatments [Count of Participants; unit: Participants]
  Radiation | 44 | 47 | 91
  Chemotherapy | 35 | 54 | 89
  Surgery | 66 | 79 | 145
  Hormone | 46 | 50 | 96
  Other | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Support Care Needs Survey (SCNS) Score
Description: The SCNS uses 57 items to measure how much help the respondent needs. Responses are given on a scale from 1 to 5 where 1 = no help is needed and 5 = high need for help. Total scores range from 57 to 285 and higher scores indicate greater need for help.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 84.15 (28.77) | 85.01 (29.44)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 79.27 (27.21) | 78.20 (23.94)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 77.20 (25.95) | 78.33 (22.71)

2. Primary Outcome: Memorial Symptom Assessment Scale-Short Form (MSAS-SF) Score
Description: Physical and psychological symptoms are assessed using the Memorial Symptom Assessment Scale-Short Form (MSAS-SF). The MSAS-SF asks if the respondent has experienced any of 32 specific symptoms during the past week, with the opportunity for the participant to enter additional symptoms. The degree of distress experienced by 28 of the symptoms is measured on a scale from 0 (not at all) to 4 (very much). The total score is the average of the responses to the distress scale items and and ranges from 0 to 4 with higher values indicating greater distress experienced from symptoms.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 1.68 (0.46) | 1.84 (0.55)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 1.71 (0.55) | 1.74 (0.41)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 1.69 (0.47) | 1.66 (0.39)

3. Primary Outcome: Functional Assessment of Cancer Therapy Scale-Breast Cancer (FACT-B) Score
Description: Quality of life is assessed using the FACT-B. The FACT-B includes 41 items which are responded to on a scale from 0 to 4, where 0 = not at all and 4 = very much. The total score ranges from 0 to 164 and higher scores indicate better quality of life.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 102.97 (21.43) | 98.72 (23.13)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 102.92 (22.14) | 103.05 (26.37)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 100.86 (22.29) | 102.03 (22.30)

4. Secondary Outcome: Questions on Attitudes, Self-Efficacy, Perceived Barriers, and Social Influences (QASPS) Score for Attitudes
Description: Attitudes related to breast cancer survivorship are measured using the Questions on Attitudes, Self-Efficacy, Perceived Barriers, and Social Influences (QASPS). The Attitudes section of this questionnaire includes 6 items scaled from -3 to 3, where -3 is the most negative score and 3 is the most positive score. There are also 7 qualitative questions. The total score for the scaled items ranges from -18 to 18 and higher scores indicate a better attitude towards breast cancer survivorship.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | -3.44 (10.82) | -0.57 (10.21)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | -3.15 (9.66) | -1.60 (9.53)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | -3.85 (9.43) | -1.76 (8.84)

5. Secondary Outcome: Questions on Attitudes, Self-Efficacy, Perceived Barriers, and Social Influences (QASPS) Score for Perceived Barriers
Description: Perceived barriers related to breast cancer survivorship are measured using the Questions on Attitudes, Self-Efficacy, Perceived Barriers, and Social Influences (QASPS). The Perceived Barriers section of this questionnaire includes 16 items where responses are given on a 4-point scale where 1 = never and 4 = always. Total scores range from 16 to 64 and higher scores indicate greater perceived barriers related to breast cancer survivorship.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 27.49 (8.45) | 30.50 (9.57)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 28.00 (8.12) | 29.48 (8.54)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 29.05 (7.97) | 28.65 (8.12)

6. Secondary Outcome: Questions on Attitudes, Self-Efficacy, Perceived Barriers, and Social Influences (QASPS) Score for Social Influences
Description: Social influences related to breast cancer survivorship are measured using the Questions on Attitudes, Self-Efficacy, Perceived Barriers, and Social Influences (QASPS). The Social Influences section of this questionnaire includes 3 items where responses are given on a 7-point scale where 1 = disapproval from social support and 7 = approval from social support. Total scores range from 3 to 21 and higher scores indicate greater positive support from social influences.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 17.12 (4.28) | 16.18 (4.18)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 17.19 (3.82) | 16.39 (4.14)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 16.32 (4.23) | 16.82 (3.71)

7. Secondary Outcome: Cancer Behavior Inventory-Brief Version (CBI-B) Score
Description: Self-efficacy related to breast cancer survivorship is measured using the Cancer Behavior Inventory-Brief Version (CBI-B). The CBI-B has 12 items assessing the degree of confidence respondents have with certain coping behaviors on a scale from 1 (not at all confident) to 9 (totally confident). Total scores range from 12 to 108 where higher scores indicate greater self-efficacy concerning cancer behaviors.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 86.04 (21.14) | 84.53 (22.00)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 89.53 (19.91) | 86.23 (18.01)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 87.22 (17.71) | 88.49 (16.52)

8. Secondary Outcome: Personal Resource Questionnaire (PRQ-2000) Score
Description: The Personal Resource Questionnaire (PRQ-2000) is a 15-item survey asking how much participants agree or disagree with statements related to social resources on a scale from 1 (strongly disagree) to 7 (strongly agree). Total scores range from 15 to 105 and higher scores indicate greater social resources.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 84.67 (13.46) | 80.01 (16.45)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 84.14 (12.99) | 80.47 (14.23)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 84.15 (11.00) | 82.17 (13.24)

9. Secondary Outcome: Perceived Isolation Scale (PIS) Score
Description: The Perceived Isolation Scale (PIS) includes 9 items asking questions about how social connectedness. Responses are rated on a 3-point scale where 1 = hardly ever, 2 = some of the time, and 3 = often. The total score is the average of the responses to the PIS items and ranges from 1 to 3 with lower scores indicating greater social connectedness.
Time Frame: Baseline, Month 1, Month 3
Population: This analysis includes participants who completed the assessment at the indicated time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | TICAA
Number analyzed (Participants) | 95 | 104
score on a scale
  Baseline | 1.61 (0.34) | 1.73 (0.47)
  Month 1: number analyzed (Participants) | 83 | 76
  Month 1 | 1.62 (0.38) | 1.70 (0.38)
  Month 3: number analyzed (Participants) | 78 | 69
  Month 3 | 1.62 (0.39) | 1.68 (0.40)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time consent to participate in the study was given through the final assessment at Month 3.
Arm/Group | Control | TICAA
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/104
Other Adverse Events (participants affected / at risk) | 0/95 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT02803593/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT02803593/ICF_001.pdf